CLINICAL TRIAL: NCT01894880
Title: Pilot Study: Sectio Bonding/Early Skin-to-skin Contact (SSC) After Caesarean Section
Acronym: SSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-425ex12/13
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Early Skin-to-skin Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early SSC (Active Comparator): Early SSC: bonding straight after birth
  Interventions: Procedure: early SSC
- late SSC (Other): late SSC: bonding after termination of operation
  Interventions: Procedure: late SSC

INTERVENTIONS:
Procedure: early SSC — bonding straight after birth
  Arms: early SSC
Procedure: late SSC — bonding after termination of operation
  Arms: late SSC

SUMMARY:
In the past decades frequency of cesarean section was increasing. Bonding or early skin-to-skin contact (SSC) starts ideally straight after birth. After vaginal delivery bonding/early SSC is already well-established. After cesarean section this important process starts after termination of operation. A Cochran review analyzed randomized studies and shows positive effects of early SSC. Possible concerns to adopt bonding in the operating room are beside organizational ones (change of established processes) also a different ambiance in the operating room (temperature, light, noise). In a prospective randomized trial, early SSC after cesarean section should be analyzed.

Hypothesis

Mothers, who have the chance to bond immediately after birth in the operating room, have lower cortisol, chromogranin A and alpha amylase levels as well as higher oxytocin levels. Adaptation of the newborn is within the normal range. Early bonding has a further positive effect on breast feeding, maternal pain processing and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* signed written informed consent
* single pregnancy
* elective cesarean section (between 7am and 15pm)
* Bleeding prophylaxis with Pabal® (carbetocin)

Exclusion Criteria:

* Age < 18 years
* disabled to give signed written informed consent
* Disease of mother or unborn, which could influence the study or makes the study impossible (e.g. severe malformation)
* Non elective cesarean
* Desire to wean
* Desire to leave the hospital within 6 hours after birth
* Bleeding prophylaxis with Syntocinon® (oxytocin)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change of oxytocin level | before, 0 min and 25 minutes after birth

SECONDARY OUTCOMES:
Change of cortisol level | before, 0 min and 25 min after birth
Change of alpha Amylase level | before, 0 min and 25 min after birth
Change of chromogranin A level | before, 0 min and 25 min after birth

OTHER OUTCOMES:
Change of pain scores on the Visual Analog Scale (VAS) | day 1 and 2 after birth
Post natal Depression (edinburgh post natal Depression scale) | day 4 after birth
Post natal Depression (edinburgh post natal Depression scale) | 6 weeks after birth
Bonding behaviour (Postpartum Bonding Questionnaire ) | day 4 after birth

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kollmann, MD, Principal Investigator — Medical University of Graz; Philipp Klaritsch, MD, Study Chair — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Graz, Austria

REFERENCES:
- [Derived] Kollmann M, Aldrian L, Scheuchenegger A, Mautner E, Herzog SA, Urlesberger B, Raggam RB, Lang U, Obermayer-Pietsch B, Klaritsch P. Early skin-to-skin contact after cesarean section: A randomized clinical pilot study. PLoS One. 2017 Feb 23;12(2):e0168783. doi: 10.1371/journal.pone.0168783. eCollection 2017. PMID 28231274